CLINICAL TRIAL: NCT00658333
Title: A Multicenter, Randomized, Double Blind, Double Dummy Controlled Study to Assess the Tolerability of an Increased Dose of Enteric Coated MPA After Conversion From MMF in Renal Transplant Recipients Who Required MMF Dose Reductions Due to Gastrointestinal Symptoms
Brief Title: A Study Designed to Compare the Tolerability of an Increased Dose of Enteric-coated Mycophenolate Acid (MPA) in Renal Transplant Patients Whose Dose of Mycophenolate Mofetil (MMF) Was Reduced Due to Gastrointestinal Symptoms
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CERL080AUS67
Record Dates: First submitted 2008-01-23; First posted 2008-04-15 (Estimated); Results first posted 2011-03-11 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-07

CONDITIONS: Renal Transplantation
Keywords: Renal Transplantation; Immunosuppression; Renal transplant recipients; Gastrointestinal symptoms associated with MMF therapy
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Enteric-coated Mycophenolate Acid (Experimental): Equimolar dose of enteric-coated mycophenolate acid with mycophenolate mofetil placebo. 1000 mg mycophenolate mofetil = 720 mg enteric-coated mycophenolate acid (MPA equivalent dose). The active and placebo study medications were dispensed in separate bottles identified as Bottle A and Bottle B.
  Interventions: Drug: Enteric-coated Mycophenolate Acid (EC-MPA); Drug: Placebo MMF
- Mycophenolate Mofetil (Active Comparator): Mycophenolate mofetil therapy with placebo enteric-coated mycophenolate acid. The active and placebo study medications were dispensed in separate bottles identified as Bottle A and Bottle B.
  Interventions: Drug: Mycophenolate Mofetil (MMF); Drug: Placebo EC-MPA

INTERVENTIONS:
Drug: Enteric-coated Mycophenolate Acid (EC-MPA)
  Other Names: myfortic®
  Arms: Enteric-coated Mycophenolate Acid
Drug: Mycophenolate Mofetil (MMF)
  Other Names: CellCept®
  Arms: Mycophenolate Mofetil
Drug: Placebo MMF
  Arms: Enteric-coated Mycophenolate Acid
Drug: Placebo EC-MPA
  Arms: Mycophenolate Mofetil

SUMMARY:
To determine if conversion to enteric coated MPA allows an escalated dose of mycophenolic acid (MPA) to be tolerated in patients experiencing gastrointestinal (GI) symptoms

ELIGIBILITY:
Inclusion criteria:

* Recipients of first or second cadaveric, living unrelated or living related kidney transplant.
* Patients on a reduced daily dose (500mg to 1500mg) of MMF with existing but tolerable and controlled gastrointestinal symptoms.
* Recipients who are at least 4 weeks post renal transplantation with stable renal function.

Exclusion criteria:

* Multi organ transplant or previous transplant with organ other than kidney
* History of GI disorder prior to transplant
* Evidence of GI disorder induced by infection, underlying medical condition, or con med other than MMF
* Modification of GI med or MMF dose within one week
* Evidence of graft rejection, treatment of acute rejection, unstable renal function within 1 week of (baseline) visit

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Novartis, Phoenix, Arizona
  - Novartis, Los Angeles, California
  - Novartis, Orange, California
  - Novartis, San Diego, California
  - Novartis, San Francisco, California
  - Novartis, Aurora, Colorado
  - Novartis, Washington D.C., District of Columbia
  - Novartis, Orlando, Florida
  - Novartis, New Orleans, Louisiana
  - Novartis, Portland, Maine
  - Novartis, Baltimore, Maryland
  - Novartis, Boston, Massachusetts
  - Novartis, Springfield, Massachusetts
  - Novarits, Detroit, Michigan
  - Novartis, New York, New York
  - Novartis, Charlotte, North Carolina
  - Novartis, Durham, North Carolina
  - Novartis, Greenville, North Carolina
  - Novartis, Winston-Salem, North Carolina
  - Novarits, Fargo, North Dakota
  - Novartis, Cleveland, Ohio
  - Novartis, Portland, Oregon
  - Novartis, Philadelphia, Pennsylvania
  - Novartis, Providence, Rhode Island
  - Novartis, Nashville, Tennessee
  - Novartis, Dallas, Texas
  - Novartis, Houston, Texas
  - Novartis, Temple, Texas
  - Novartis, Murray, Utah
  - Novartis, Burlington, Vermont
  - Novartis, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in the US from March 2008 to March 2009.
Pre-assignment Details: Patients were screened for eligibility. If eligible, willing to participate and provided informed consent, patients were randomized in a blinded fashion to either an equimolar dose of enteric-coated mycophenolate acid (MPA) or remained on the current dose of mycophenolate mofetil (MMF).
Period: Overall Study
Arm/Group | Enteric-coated Mycophenolate Acid | Mycophenolate Mofetil
Started | 15 | 15
Completed | 13 | 14
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enteric-coated Mycophenolate Acid | Mycophenolate Mofetil | Total
Number analyzed (Participants) | 15 | 15 | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 51.3 (12.54) | 49.8 (12.45) | 50.5 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response (Yes/no)
Description: The primary variable was the response (yes/no) with positive response being defined as an increase of 360 mg/day enteric-coated mycophenolate acid (MPA)from the baseline daily dose, tolerated and maintained for a 4 week duration until the end of the study (Week 6). Tolerability was defined as the overall assessment of improvement or no change in the intensity of physician assessed gastrointestinal (GI) symptoms at end of study as reported on the physician administered evaluation of GI symptomatology.
Time Frame: 6 weeks
Population: Intent to Treat Population
Measure: Number; unit: Participants
Arm/Group | Enteric-coated Mycophenolate Acid | Mycophenolate Mofetil
Number analyzed (Participants) | 15 | 15
Participants
  Yes | 10 | 9
  No | 5 | 6

2. Secondary Outcome: Average Daily Doses (mg) of Enteric-coated Mycophenolate Acid (MPA) and Mycophenolate Mofetil (MMF) by Treatment Duration Intervals
Description: The average daily doses of enteric-coated mycophenolate acid (MPA) and mycophenolate mofetil (MMF) at baseline and during the last 2 weeks of treatment. 1000 mg MMF = 720 mg enteric-coated MPA (MPA equivalent dose).
Time Frame: Baseline and week 4 to week 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Enteric-coated Mycophenolate Acid | Mycophenolate Mofetil
Number analyzed (Participants) | 15 | 15
mg
  MMF Baseline Dose (n=15, 15) | 1033.30 (351.87) | 1216.7 (364.33)
  Week 4 to Week 6 (n=13, 14) | 914.5 (419.85) | 1567.6 (442.55)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Safety population
Arm/Group | Enteric-coated Mycophenolate Acid | Mycophenolate Mofetil
Serious Adverse Events (participants affected / at risk) | 2/15 | 0/15
Other Adverse Events (participants affected / at risk) | 12/15 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enteric-coated Mycophenolate Acid (N=15) | Mycophenolate Mofetil (N=15)
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enteric-coated Mycophenolate Acid (N=15) | Mycophenolate Mofetil (N=15)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 3
Defaecation urgency (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 4
Eructation (Gastrointestinal disorders) | 2 | 3
Flatulence (Gastrointestinal disorders) | 3 | 4
Gastrointestinal disorder (Gastrointestinal disorders) | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 4
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Human polyomavirus infection (Infections and infestations) | 1 | 0
Sputum purulent (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Complications of transplant surgery (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Eosinophil count increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 1
Weight increased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to the insufficient number of patients enrolled in the study, no conclusions can be made from the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.